CLINICAL TRIAL: NCT00028314
Title: A Restrictively Randomized, Open-Label, Controlled, Pilot Study of the Effect of a Thymidine Analogue Substitution or Change to a Nucleoside-Sparing Regimen on Peripheral Fat Wasting
Brief Title: Effects of Treatment Changes on Fat Wasting in the Arms and Legs of HIV Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: A5110; AACTG A5110; ACTG A5110
Record Dates: First submitted 2001-12-20; First posted 2001-12-21 (Estimated); Last update posted 2013-07-29 (Estimated); Status verified 2013-07

CONDITIONS: HIV Infections; Lipodystrophy; Wasting Disease
Keywords: HIV-1; Abacavir; Nevirapine; Ritonavir; RNA, Viral; HIV Protease Inhibitors; Reverse Transcriptase Inhibitors; Anti-HIV Agents; Viral Load; HIV Wasting Syndrome; ABT 378; Treatment Experienced
MeSH Terms: conditions — HIV Infections; Lipodystrophy; Wasting Syndrome; HIV Wasting Syndrome | interventions — abacavir; atazanavir, ritonavir drug combination; Lopinavir; Nevirapine

INTERVENTIONS:
Drug: Abacavir sulfate
Drug: Atazanavir/Ritonavir
Drug: Lopinavir/Ritonavir
Drug: Nevirapine

SUMMARY:
The goals of this study are to find out if fat wasting and weight loss in the arms and legs of HIV patients taking highly active antiretroviral therapy (HAART) are caused by nucleoside/nucleotide reverse transcriptase inhibitors (NRTIs) and if wasting can be reversed if the NRTI is stopped and replaced with other anti-HIV drugs.

DETAILED DESCRIPTION:
Recent studies suggest body shape changes, fat redistribution, and fat lipoatrophy may be related to the NRTI component of patients' HAART and not to the protease inhibitor (PI) component. The hypothesis of this study is that thymidine analogues such as stavudine (d4T) and zidovudine (ZDV) cause lipoatrophy more so than non-thymidine analogues and that removal of thymidine analogues from HAART in patients with defined lipoatrophy will reverse this process.

In Step 1, patients will undergo axial mid-thigh and abdomen computer tomography (CT) scans. If the CT scans are readable, patients are restrictively and randomly assigned to 1 of 2 treatment arms in Step 2. Patients in Arm A-1 will replace the thymidine analogue component (stavudine [d4T] or zidovudine [ZDV]) of their HAART with abacavir (ABC). Patients in Arm B-1 will discontinue their current HAART and will receive a PI and a nonnucleoside reverse transcriptase inhibitor (NNRTI), either lopinavir/ritonavir (LPV/r) and nevirapine (NVP) or atazanavir, ritonavir, and NVP. Patients currently on efavirenz (EFV) not provided by the study may choose to continue with EFV instead of switching to NVP. Comparisons will be made to the baseline values of subcutaneous fat measured by mid-thigh and abdominal CT. Patients in Arms A-1 and B-1 remain on study for a total of 48 weeks and do not advance to Step 3.

Two additional groups (Arms A-2 and B-2) made no changes to HAART for 28 weeks to evaluate the natural history of change in lipoatrophy over time; accrual into these groups and into Step 3 has been discontinued. At Week 28, patients in Arms A-2 and B-2 were registered to Step 3 and switched from HAART to a designated new treatment. Arm A-2 patients will replace d4T or ZDV with ABC for 48 weeks. Arm B-2 patients replace their HAART with LPV/r plus NVP for 48 weeks. If patients in Arms A-2 and B-2 have not completed the 28-week delay and have not switched regimens, they will enter Step 4 and be reregistered into Arms A-1 and B-1, respectively, remaining on their treatment assignment for 48 weeks. If patients in Arms A-2 and B-2 have already switched regimens, then they will continue on their new regimens until Week 76.

ELIGIBILITY:
Note: accrual into Arms A-2 and B-2 of this study has been discontinued.

Inclusion Criteria for Step 1

* HIV infected
* Experiencing a loss of fat since starting anti-HIV therapy, especially in the arms and legs
* Receiving anti-HIV therapy of 3 or more drugs, including either stavudine or zidovudine, for 24 weeks or more prior to study screening
* Viral load less than 500 copies/ml at study screening and within 60 days prior to study entry
* CD4 count of 100 or more cells/mm3 obtained within 60 days prior to study entry
* Approved methods of contraception
* Written informed consent

Exclusion Criteria for Step 1

* Currently receiving abacavir sulfate or have received abacavir sulfate in the past AND any or all of the following: unable to tolerate lopinavir/ritonavir (LPV/r) or nevirapine (NVP); failed anti-HIV treatment containing LPV/r, any other 2 PIs, or any other NNRTI; taking lamivudine (3TC) or tenofovir disoproxil fumarate (TDF) for hepatitis B virus infection and need to remain on a 3TC- or TDF-containing regimen; or have a low chance of response to LPV/r plus NVP
* Cancer treatment 6 months prior to study entry
* Initiated oral drugs to lower blood sugar level 24 weeks prior to study entry. Patients who have taken oral drugs to lower their blood sugar levels for 24 weeks or more prior to study entry are eligible.
* Began therapy with male sex hormones 24 weeks prior to study entry. Patients who have had continuous, stable therapy with male sex hormones for 24 weeks or more prior to study entry are eligible.
* Certain medications within 14 days prior to study entry
* Serious illness within 14 days prior to study entry
* Hepatitis within 60 days prior to study entry
* Thyroid problems
* Drug or alcohol use which, in the opinion of the investigator, would interfere with the study
* Currently using experimental agents except when approved by the study
* Pregnant or breastfeeding

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 150
Dates: Start 2002-03; Study Completion 2005-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert L Murphy, MD, Study Chair — Northwestern University Medical Center; Pablo Tebas, MD, Study Chair — University of Pennsylvania, Adult Clinical Trials Unit
Locations (25):
- United States (25):
  - UCLA CARE Center CRS, Los Angeles, California
  - Harbor-UCLA Med. Ctr. CRS, Torrance, California
  - University of Colorado Hospital CRS, Aurora, Colorado
  - Univ. of Hawaii at Manoa, Leahi Hosp., Honolulu, Hawaii
  - Northwestern University CRS, Chicago, Illinois
  - Rush Univ. Med. Ctr. ACTG CRS, Chicago, Illinois
  - Cook County Hosp. CORE Ctr., Chicago, Illinois
  - Indiana Univ. School of Medicine, Infectious Disease Research Clinic, Indianapolis, Indiana
  - Indiana Univ. School of Medicine, Wishard Memorial, Indianapolis, Indiana
  - Methodist Hosp. of Indiana, Indianapolis, Indiana
  - Beth Israel Deaconess Med. Ctr., ACTG CRS, Boston, Massachusetts
  - SSTAR, Family Healthcare Ctr., Fall River, Massachusetts
  - University of Minnesota, ACTU, Minneapolis, Minnesota
  - St. Louis ConnectCare, Infectious Diseases Clinic, St Louis, Missouri
  - Washington U CRS, St Louis, Missouri
  - Beth Israel Med. Ctr., ACTU, New York, New York
  - NY Univ. HIV/AIDS CRS, New York, New York
  - Univ. of Cincinnati CRS, Cincinnati, Ohio
  - MetroHealth CRS, Cleveland, Ohio
  - The Ohio State University Medical Center, Columbus, Ohio
  - Hosp. of the Univ. of Pennsylvania CRS, Philadelphia, Pennsylvania
  - The Miriam Hosp. ACTG CRS, Providence, Rhode Island
  - Rhode Island Hosp., Providence, Rhode Island
  - Vanderbilt Therapeutics CRS, Nashville, Tennessee
  - Univ. of Texas Medical Branch, ACTU, Galveston, Texas

REFERENCES:
- [Background] Calza L, Manfredi R, Chiodo F. Dyslipidaemia associated with antiretroviral therapy in HIV-infected patients. J Antimicrob Chemother. 2004 Jan;53(1):10-4. doi: 10.1093/jac/dkh013. Epub 2003 Nov 25. PMID 14645323
- [Background] Calza L, Manfredi R, Chiodo F. Hyperlipidaemia in patients with HIV-1 infection receiving highly active antiretroviral therapy: epidemiology, pathogenesis, clinical course and management. Int J Antimicrob Agents. 2003 Aug;22(2):89-99. doi: 10.1016/s0924-8579(03)00115-8. PMID 12927947
- [Background] Carr A, Miller J, Law M, Cooper DA. A syndrome of lipoatrophy, lactic acidaemia and liver dysfunction associated with HIV nucleoside analogue therapy: contribution to protease inhibitor-related lipodystrophy syndrome. AIDS. 2000 Feb 18;14(3):F25-32. doi: 10.1097/00002030-200002180-00001. PMID 10716495
- [Background] McComsey G. Update on mitochondrial toxicity of antiretrovirals and its link to lipodystrophy. AIDS Rev. 2002 Jul-Sep;4(3):140-7. PMID 12416448
- [Background] Mallal SA, John M, Moore CB, James IR, McKinnon EJ. Contribution of nucleoside analogue reverse transcriptase inhibitors to subcutaneous fat wasting in patients with HIV infection. AIDS. 2000 Jul 7;14(10):1309-16. doi: 10.1097/00002030-200007070-00002. PMID 10930144
- [Result] Tebas P, Zhang J, Hafner R, Tashima K, Shevitz A, Yarasheski K, Berzins B, Owens S, Forand J, Evans S, Murphy R. Peripheral and visceral fat changes following a treatment switch to a non-thymidine analogue or a nucleoside-sparing regimen in HIV-infected subjects with peripheral lipoatrophy: results of ACTG A5110. J Antimicrob Chemother. 2009 May;63(5):998-1005. doi: 10.1093/jac/dkp071. Epub 2009 Mar 19. PMID 19299471